CLINICAL TRIAL: NCT06462365
Title: Phase I, First in Human, Open Label Study to Evaluate Safety and Tolerability of TRX103 Cells in Subjects With Hematological Malignancies Undergoing HLA-mismatched Related or Unrelated Hematopoietic Stem Cell Transplantation (HSCT)
Brief Title: Prevention of GvHD in Participants With Hematological Malignancies Undergoing Hematopoietic Stem Cell Transplant (HSCT)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Tr1X, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: TRX103-01
Record Dates: First submitted 2024-06-06; First posted 2024-06-17 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2024-10

CONDITIONS: Hematologic Malignancy; GvHD; GVHD,Acute; GVHD, Chronic; Hematopoietic Stem Cell Transplant; Acute Lymphoblastic Leukemia, Adult B-Cell; Acute Lymphoblastic Leukemia, Adult T-Cell; Acute Myeloid Leukemia in Remission; Myelodysplastic Syndromes; Chronic Myelomonocytic Leukemia, in Remission; Cancer Remission
Keywords: AML; CMML; Stem Cell Transplant; B-ALL; T-ALL; Acute GvHD; Graft versus Host Disease; Chronic GvHD; MDS; Cellular Therapy; Autoimmune; T regulatory cells
MeSH Terms: conditions — Hematologic Neoplasms; Bronchiolitis Obliterans Syndrome; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Graft vs Host Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- TRX-103 (Experimental): TRX-103 will be infused on time post hematopoietic stem cell transplant (HSCT).
  Interventions: Biological: TRX103

INTERVENTIONS:
Biological: TRX103 — TRX103 infusion via central line.

SUMMARY:
The purpose of this Phase 1, first in human open-label study is to assess the safety and tolerability of TRX-103 in patients with hematological malignancies undergoing HLA-mismatched related or unrelated hematopoietic stem cell transplantation (HSCT). It is anticipated that up to 36 Subjects will be enrolled during a 18-24 month enrollment period. TRX-103 will be infused one time post HSCT.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with one of the following hematologic malignancies: Acute Lymphoblastic Leukemia (B- or T-ALL), Acute Myeloid Leukemia (AML) and Myelodysplastic Syndrome (MDS), or Chronic myelomonocytic leukemia (CMML)
2. Males and Females Age ≥ 18 years.
3. Weight of ≥ 35 Kg.
4. Karnofsky performance status ≥ 70 %.
5. Available mismatched related (haploidentical) or unrelated donors for peripheral blood stem cell (PBSC) donation.
6. Subjects must otherwise fulfill institutional criteria for eligibility to undergo allogeneic stem cell transplantation.
7. Absence of uncontrolled bacterial, viral or fungal infection at time of enrollment.
8. Have adequate organ function.
9. Subjects > 65-year-old receiving MAC conditioning will only be eligible if they have a HSCT-comorbidity index score < 5.
10. Subjects must be able to understand and sign informed consent and be willing and able to complete all specified procedures and visits.

Exclusion Criteria:

1. Prior allogeneic bone marrow, peripheral blood, or cord blood HSCT.
2. Any subject with a history of significant renal, hepatic, pulmonary, or cardiac dysfunction, or on treatment to support cardiac dysfunction.
3. HIV positive.
4. Positive hepatitis-B surface antigen. Subject may be included if they are HBV PCR negative.
5. Positive hepatitis-C antibody with positive Recombinant Immunoblot Assay (RIBA) or PCR unless the subject has received curative anti-viral treatment and confirmed negative viral load by PCR.
6. Received another investigational agent for treatment of disease understudy within 28 days (or 5 half-lives, whichever is shorter) of conditioning and/or have not recovered from treatment related toxicities.
7. Subjects with a previous history of Thrombotic Thrombocytopenic Purpura (TTP) or Hemolytic Uremic Syndrome (HUS) who are not good candidates for treatment with sirolimus.
8. Subjects that are pregnant, breast feeding or aim to become pregnant during the study period. (Subjects must agree to use a highly effective method of contraception).
9. Any serious illness, uncontrolled inter-current illness, psychiatric illness, active or uncontrolled infection, or other medical condition or history, including laboratory results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-04-08 (Actual); Primary Completion 2026-04-15 (Estimated); Study Completion 2027-04-15 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of TRX103 cell infusion through incidence of Adverse events. | Up to a year
Safety of TRX103 determined by stem cell engraftment and donor chimerism after HSCT measured by absolute neutrophil counts and percent donor chimerism. | Up to day 42
Safety of TRX103 determined by negative Replication Competent Lentivirus (RCL). | At 3-month, 6-month, and 1-year.

SECONDARY OUTCOMES:
Incidence of Grade II-IV acute GvHD (aGvHD). | Day 0 to Day +100 day
Incidence of Grade III-IV acute GvHD (aGvHD). | Day 0 to Day +100 day
Incidence and severity of chronic GvHD (cGvHD) | Day +100 through Day +365
Overall survival at Day +365. | Up to a year

CONTACTS AND LOCATIONS:
Overall Officials: Maria Grazia Roncarolo, MD, Study Director — Tr1X, Inc.
Locations (5):
- United States (5):
  - City of Hope, Duarte, California
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Fred Hutchinson Cancer Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No